CLINICAL TRIAL: NCT04808596
Title: Pulmonary Hypertension Biorepository and Registry
Acronym: PHBR
Status: Recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Leslie Spikes, MD, Associate Professor, University of Kansas Medical Center
Other Study IDs: STUDY#00145817
Record Dates: First submitted 2021-03-17; First posted 2021-03-22 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Hypertension; Pulmonary Arterial Hypertension; Pulmonary Hypertension Due to Left Heart Disease; Pulmonary Hypertension, Primary; Pulmonary Hypertension Due to Lung Diseases and Hypoxia; Pulmonary Hypertension, Primary, 4; Pulmonary Hypertension, Primary, 2; Pulmonary Hypertension, Primary, 3; Chronic Thromboembolic Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension; Familial Primary Pulmonary Hypertension; Hypoxia; Lipodystrophy, Congenital Generalized, Type 3

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Future projects might include genetic testing on your samples. Genetic testing studies pieces of DNA called genes. The cells in your body contain deoxyribonucleic acid, or DNA for short. DNA is passed down from your parents. It carries the genes that determine how you look and how your body works and tells a genetic story about you. Differences in genes may help explain why a particular drug is effective and safe in some people, but not in others. Differences in genes also may explain why some people get certain diseases, but others do not. The genetic information may be important in guiding targeted treatments in the future.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Establish a pulmonary hypertension registry and biorepository to lead towards a further understanding of the disease.

DETAILED DESCRIPTION:
The aim of this project will be to establish a broad and wide-ranging registry and biorepository of blood samples from patients with pulmonary hypertension, including all WHO groups I-V to be used for future research in these areas. This will be both a retrospective and prospective project. The registry and biorepository will be utilized to study and grow our knowledge of the cellular mechanisms and mediators of the disease and, in turn, contribute to advancements in treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is a patient at TUKHS or has agreed to participate in a study approved by the KUMC Human Research Protection Program (HRPP)
2. The participant has a diagnosis of pulmonary hypertension confirmed by right heart catheterization
3. Patient is ≥ 18 years of age or older

Exclusion Criteria:

1. Participant declines to participate (living patients only)
2. Participant is unable to provide informed consent (living patients only)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Pulmonary Hypertension Group 1-5
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-08-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Collect Clinical Data | From Enrollment to 6 Months
  Collect clinically obtained data from current and deceased patients with pulmonary hypertension to support research.
Establish a Biorepository | From Enrollment to 6 Months
  Establish a collection of biospecimens from patients with pulmonary hypertension.
Biospecimens Collection | From Enrollment to 12 Months
  Correlate biospecimens to longitudinally collected individual patient data.
Collaborate | From Enrollment to 24 Months
  Provide biospecimens to researchers investigating pulmonary hypertension. Separate IRB approval will be needed for these studies.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie A Spikes, MD, Principal Investigator — Assistant Professor of Medicine; Luigi R Boccardi, Ed.D., MPH, Study Director — Director of Pulmonary Research
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Contact Luigi Boccardi to discuss accessing IPD.